CLINICAL TRIAL: NCT07379541
Title: Effects of Mindfulness-of-Death Meditation on Problematic Smartphone Use in Emerging Adulthood
Brief Title: Meditation-Based Online Psychological Intervention: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, li,xinyi, Co-Investigator, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BNU-poslab-MLD-2025
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Smartphone Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Meditation Intervention Group (Experimental): A 16-day mindfulness-based curriculum was implemented as the intervention, with participants completing one 20-min session daily via the online platform.
  Interventions: Behavioral: Mindful Breathing Practice (MBP) - 16-Day Online Meditation Course
- Mindfulness-of-Death Group (Experimental): A 16-day mindfulness-of-death curriculum was implemented as the intervention, with participants completing one 20 min online session daily.
  Interventions: Behavioral: Mindfulness of Death (MoD) - 16-Day Online Meditation Course
- Wait-list Control Group (No Intervention): Wait-list Control Group

INTERVENTIONS:
Behavioral: Mindfulness of Death (MoD) - 16-Day Online Meditation Course — The Mindfulness of Death (MoD) intervention is a 16-day online meditation program designed to cultivate awareness of death. The course consists of 16 daily sessions (approximately 20 minutes each), including brief psychoeducational content and guided meditation practice. The initial sessions focus on breathing-based mindfulness to establish attentional stability, followed by mindfulness of death practices that emphasize the inevitability and uncertainty of death while encouraging attention to life and the present moment. The intervention adopts a non-religious approach and does not require participants to hold any religious or spiritual beliefs.
  Arms: Mindfulness-of-Death Group
Behavioral: Mindful Breathing Practice (MBP) - 16-Day Online Meditation Course — The Mindful Breathing Practice (MBP) intervention is a 16-day online meditation program designed to cultivate present-moment awareness by intentionally anchoring attention on the natural rhythm of breathing. The course consists of 16 daily sessions (approximately 15 minutes each), including brief instructional guidance and guided mindful breathing exercises. Participants are guided to observe the bodily sensations of inhalation and exhalation (e.g., the airflow at the nostrils or the rise and fall of the abdomen) and, when attention wanders, to gently bring it back to the breath with a non-judgmental and accepting attitude. The intervention adopts a non-religious approach, involves no spiritual or religious content, and is suitable for the general population.
  Arms: Mindfulness-Meditation Intervention Group

SUMMARY:
relationships. As the primary users of smartphones, emerging adults represent a key population for such research. Using a randomised controlled trial, we compared mindfulness-of-death meditation with traditional mindfulness meditation to evaluate the unique effects of the former on problematic smartphone use. We also examined potential psychological pathways-namely increases in self-esteem and meaning in life, and reductions in perceived stress-through which the intervention may exert its benefits.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were adults aged 18-29 years who:

* reported no current or past psychiatric diagnosis,
* exhibited problematic smartphone use,
* and had a mean daily screen-on time exceeding four hours.
* Exclusion criteria were as follows:
* aged <18 or ≥30 years;
* any current or past psychiatric diagnosis;
* self-reported absence of problematic smartphone use;
* mean daily smartphone use ≤4 hours;
* currently enrolled in any meditation-based intervention;
* use of psychoactive medication or concurrent psychological treatment;
* participation in another psychological intervention trial.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2025-02-23 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' problematic smartphone use was assessed using the 33-item Smartphone Addiction Scale (SAS) [Kwon et al., 2013]. Although the original scale employed a 6-point response format, the present study utilized a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always; α = .88). The scale comprises six dimensions: daily disturbance, positive anticipation, withdrawal symptoms, online intimacy, excessive use, and tolerance. Higher total scores indicate greater severity of problematic smartphone use.

SECONDARY OUTCOMES:
Perceived Stress Scale-10 | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' perceived stress was assessed using the 10-item Perceived Stress Scale (PSS-10) [Cohen et al., 1983; Chen et al., 2021]. The validated Chinese version [Chen, Tian, Zhang, et al., 2021] was employed in the present study. Items were rated on a 5-point Likert scale ranging from 1 (never) to 5 (always; α = .78-.91). The scale consists of two dimensions: perceived helplessness and self-efficacy belief. Six items assessing self-efficacy belief were reverse-scored. Higher total scores reflect elevated levels of perceived stress.
Philadelphia Mindfulness Scale | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' mindfulness was assessed using the 10-item Philadelphia Mindfulness Scale (PHLMS) [Cardaciotto et al., 2008; Zeng et al., 2015]. The validated Chinese version [Zeng, Li, Zhang, & Liu, 2015] was employed in the present study. Items were rated on a 5-point Likert scale ranging from 1 (never) to 5 (always; awareness subscale α = .82; acceptance/avoidance subscale α = .80). The scale comprises two dimensions: awareness and acceptance/avoidance. Five items assessing acceptance/avoidance were reverse-scored. Higher total scores indicate greater mindfulness.
Self-Control Scale for College Students | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' self-control was assessed using the 19-item Self-Control Scale for College Students [Tangney et al., 2004; Tan & Guo, 2008]. The validated Chinese version [Tan & Guo, 2008] was employed in the present study. Items were rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very much; α = .85). The scale comprises five dimensions: impulse control, health habits, resisting temptation, focused work, and moderation in entertainment. Higher total scores reflect greater self-control.
Boredom Proneness Scale-Short Form | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' boredom proneness was assessed using the 12-item Short Form of the Boredom Proneness Scale (BPS-SF) [Vodanovich et al., 2005]. Items were rated on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree; external stimulation deficiency α = .81; internal stimulation deficiency α = .78). The scale comprises two dimensions: external stimulation deficiency and internal stimulation deficiency. Six items assessing internal stimulation deficiency were reverse-scored. Higher total scores indicate greater boredom proneness.
Three-Dimensional Meaning in Life Scale | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' meaning in life was assessed using the 11-item Three-Dimensional Meaning in Life Scale (3DM) [Martela & Steger, 2016]. Items were rated on a 7-point Likert scale ranging from 1 (not at all) to 7 (very much; purpose α = .90; coherence α = .84; significance α = .86). The scale comprises three dimensions: purpose, coherence, and significance. Higher total scores reflect greater meaning in life.
Zimbardo Time Perspective Inventory | Baseline, post-intervention (Day 16), and one-month follow-up
  Participants' time perspective was assessed using the 25-item Zimbardo Time Perspective Inventory (ZTPI) [Zimbardo & Boyd, 1999]. Items were rated on a 5-point Likert scale ranging from 1 (very uncharacteristic) to 5 (very characteristic; past-positive α = .79; past-negative α = .82; present-hedonistic α = .84; present-fatalistic α = .74; future α = .84). The scale comprises five dimensions: past-positive, past-negative, present-hedonistic, present-fatalistic, and future. Higher subscale scores indicate stronger orientation toward that particular time perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding sharing individual participant data (IPD) has not yet been finalized. Data may be shared in de-identified form after publication, depending on ethical approval and institutional policies at that time.